CLINICAL TRIAL: NCT01741727
Title: A Phase 1/2 Study Evaluating the Safety, Pharmacokinetics and Efficacy of ABT-414 in Subjects With Advanced Solid Tumors Likely to Over-Express the Epidermal Growth Factor Receptor (EGFR)
Brief Title: A Study of ABT-414 in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-379
Record Dates: First submitted 2012-09-19; First posted 2012-12-05 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2016-02

CONDITIONS: Squamous Cell Tumors
MeSH Terms: interventions — ABT-414

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABT-414 (Experimental): Subjects with solid tumors (Phase 1) and squamous non-small cell lung cancer (NSCLC) (Phase 2)
  Interventions: Drug: ABT-414

INTERVENTIONS:
Drug: ABT-414 — ABT-414 will be administered by intravenous infusion.

SUMMARY:
A study of ABT-414 in subjects with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a solid tumor type likely to over-express Epidermal Growth Factor Receptor (EGFR) (Phase 1)
2. Subjects have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
3. Subjects have available tumor tissue
4. Subjects have adequate bone marrow, renal, and hepatic function as follows: Bone marrow: Absolute neutrophil count (ANC) >/= 1,500/mm3 Platelets >/= 100,000/mm3; Hemoglobin >/= 9.0 g/dL Renal function: Serum creatinine </= 1.5 times the upper limit of the institution's normal range Hepatic function: Bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) </= 1.5 times the upper limit of the institution's normal range. Subjects with liver metastasis may have an AST and ALT of </= 5.0 x the upper limit of normal.
5. Subjects in the Phase 2 portion must have squamous cell Non-Small Cell Lung Cancer (NSCLC)
6. Eligibility is restricted to subjects with confirmed EGFR amplification in the EGFR amplified cohort

Exclusion Criteria:

1. The subject has uncontrolled metastases to the central nervous system (CNS). Subjects with brain metastases are eligible provided they have shown clinical and radiographic stable disease for at least 28 days after definitive therapy and have not received prior whole brain radiation (Phase 1 only).
2. The subject has received anticancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal, biologic, or any investigational therapy within a period of 28 days prior to the first dose of ABT-414.
3. The subject has unresolved clinically significant toxicities from prior anticancer therapy, defined as any Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or higher.
4. The subject had had major surgery within 28 days prior to the first dose of ABT-414.
5. The subject has a history of immunologic reaction to any Immunoglobulin G (IgG) containing agent.
6. Phase 2 portion only: The subject has previous or concurrent cancer that is distinct in primary site or histology from NSCLC, except cervical carcinoma in situ, non-melanoma carcinoma of the skin or in situ carcinoma of the bladder. Any cancer curatively treated greater than 3 years prior to entry is permitted.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Phase 1 - Safety (Number of subjects with adverse events and/or dose limiting toxicities) | Every 1-3 weeks for an average of 20 weeks
  Evaluation of vital signs, clinical lab testing, adverse event monitoring, physical exam and electrocardiogram (ECG) (periodic) under different dosing schedules, drug infusion times, and manufacturing processes.
Phase 1 - Pharmacokinetic profile | Multiple timepoints Week 1 and Week 7
  Cmax, Cmin, and half-life
Phase 2 - Efficacy | Every 6-9 weeks for an average of 20 weeks
  Objective response per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST)

SECONDARY OUTCOMES:
Phase 2- Safety (Scheduled study visits occurring on average every 3 weeks) | Followed on average every 3 weeks for approximately 20 weeks
  Evaluation of vital signs, clinical lab testing, and adverse event monitoring, physical exam, and electrocardiogram (periodic)
Phase 2- Pharmacokinetic profile | Multiple timepoints Week 1
  Cmax, Cmin, and half-life
Phase 1&2 - QT assessment | Week 1
  Triplicate electrocardiograms

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ocampo, MD, Study Director — AbbVie
Locations (6):
- United States (5):
  - Site Reference ID/Investigator# 90333, Scottsdale, Arizona
  - Site Reference ID/Investigator# 83156, Chicago, Illinois
  - Site Reference ID/Investigator# 117516, Boston, Massachusetts
  - Site Reference ID/Investigator# 83154, Boston, Massachusetts
  - Site Reference ID/Investigator# 83155, San Antonio, Texas
- Site Reference ID/Investigator# 89035, Ottawa, Canada

REFERENCES:
- [Result] Munasinghe WP, Mittapalli RK, Li H, Hoffman DM, Holen KD, Menon RM, Xiong H. Evaluation of the effect of the EGFR antibody-drug conjugate ABT-414 on QT interval prolongation in patients with advanced solid tumors likely to over-express EGFR. Cancer Chemother Pharmacol. 2017 May;79(5):915-922. doi: 10.1007/s00280-017-3284-y. Epub 2017 Mar 27. PMID 28349167